CLINICAL TRIAL: NCT06300164
Title: The Effect of Unripe Carob Fruit on Oxidative Markers and Intestinal Permeability and Microbiota in Celiac Patients
Brief Title: The Effect of Unripe Carob Fruit in Celiac Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Toros University (Other)
Responsible Party: Principal Investigator, Özlem ÖZPAK AKKUŞ, Asst.Prof., Toros University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Unripecarobinceliac
Record Dates: First submitted 2024-02-19; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Celiac Disease
Keywords: Celiac; Unripe carob; Antioxidant; Microbiota
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Intervention Model Description: The study will conduct by using a prospective randomized double-blind clinical trial model.
Who Masked: Participant, Care Provider
Masking Description: Participants will not know which type of cookies to eat.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- People with celiac disease who eat cookies with unripe carob - Experimental Group (Experimental): Individuals with celiac disease who met the inclusion criteria and participated in the study will divided into two groups by Specialist OrhN SEZGİN, and they will be asked to consume the cookies produced (in the preliminary study) produced as a standard (n=15) and with the addition of unripe carob (n=15) for eight weeks.
  The individuals participating in the study will be asked not to change their eating habits, physical activity habits, and drug treatments during the study period. Each individual participating in the study will be provided with the required amount of cookie during the study and will be contacted weekly by Ecem GÜLÜŞEN, a dietitian, to verify whether they consume cookies regularly.
  Interventions: Dietary Supplement: Unripre Carob
- No intervention - Control Group (No Intervention): Individuals with celiac disease will not eat unripe carob cookie

INTERVENTIONS:
Dietary Supplement: Unripre Carob — The standard cookies and test cookies (with carob addition) to be used in the study will be produced by Dr. Lecturer Özlem ÖZPAK AKKUŞ at Toros University Nutrition Principles Laboratory. Prof. Dr. Özlem ÖZPAK AKKUŞ will produce the cookies. For standard cookies, 1 egg, 325 g gluten-free flour (Söke flour), 75 grams butter, 50 grams sugar, 10 grams baking powder, 10 grams vanilla will be added and the prepared bread mixture will be divided into 50 equal parts. To make cookies with the addition of unripe carob, the same recipe as the standard cookie will be used to make the test cookie with the addition of unripe carob fruit flour, divided into 50 equal parts, and the amount of unripe carob fruit flour will be added by calculating the daily fiber consumption amount of the patients participating in the study to be 25 g.
  Arms: People with celiac disease who eat cookies with unripe carob - Experimental Group

SUMMARY:
The aim of this study was to investigate the effects of the consumption of cookies produced by adding the unripe part of carob fruit, which has high insoluble fiber, polyphenol and antioxidant content, on the oxidative parameters (TAS and MDA), intestinal permeability (zonulin, GIP) and microbiota of celiac patients and to develop new products containing unripe carob fruit for celiac patients in this direction.

DETAILED DESCRIPTION:
Between 01.02.2022 and 30.05.2022 by Specialist Dr. Orhan SEZGİN

The study will be conducted with 30 volunteers who present to the Mersin University Faculty of Medicine Hospital Gastroenterology Department in Mersin.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with celiac disease within a maximum period of 1 year,
* Have not received dietary treatment by a dietitian before
* Body Mass Index value between 18.5-25.0 kg/m2,
* Who have consumed carob fruit and have not had any allergies,
* Signed the Informed Consent Form,
* Between the ages of 19 and 64,
* Who has not had gastrointestinal tract surgery,
* Without mental disorder,
* Without inflammatory disease,
* No antibiotics or probiotics for the last 1 month,
* Not taking prescription drugs and/or fiber supplements,
* Not taking vitamin, mineral supplements,
* Not during pregnancy and lactation,
* Without excessive alcohol consumption (>2 drinks/day)

Exclusion Criteria:

* Diagnosed with celiac disease for more than 1 year,
* Have gastrointestinal diseases other than celiac disease,
* Have previously received dietary treatment by a dietitian, following a diet other than a gluten-free diet,
* Body Mass Index values below 18.5 kg/m2 and above 25.0 kg/m2,
* Who have consumed carob fruit and have had any allergies,
* Not signing the Informed Volunteer Consent Form,
* Not between the ages of 19-64,
* Gastrointestinal tract surgery,
* With a mental disorder,
* With inflammatory disease,
* Taking antibiotics or probiotics for the last 1 month,
* Taking prescription medication and/or fiber supplements,
* Taking vitamin and mineral supplements,
* During pregnancy and lactation,
* Excessive alcohol consumption (>2 drinks/day)

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Examination of between group differences regarding serum Total Antioxidant Capacity (TAC) | First day at the beginning of the study
  Examination of intergroup differences of the concentration of the serum total antioxidant capacity for the determination of antioxidant capacity status in celiac diseases
Examination of between group differences regarding serum Malondialdehyde (MDA) | First day at the beginning of the study
  Examination of intergroup differences of the concentration of the serum malondialdehyde for the determination of oxidant capacity status in celiac diseases
Examination of between group differences regarding serum zonulin | First day at the beginning of the study
  Examination of intergroup differences of the concentration of the serum zonulin for the determination of intestinal permeability in celiac diseases

SECONDARY OUTCOMES:
Comparison of between group differences regarding serum Total Antioxidant Capacity (TAC) | Eight weeks after the start of the study
  Comparison of between group differences of the concentration of the serum total antioxidant for the determination of antioxidant capacity status in celiac diseases
Comparison of between group differences regarding serum Malondialdehyde (MDA) | Eight weeks after the start of the study
  Comparison of between group differences of the concentration of the serum malondialdehyde for the determination of oxidant capacity status in celiac diseases
Comparison of between group differences regarding serum zonulin | Eight weeks after the start of the study
  Comparison of between group differences of the concentration of the serum zonulin for the determination of intestinal permeability in celiac diseases

IPD SHARING:
Plan to Share IPD: Yes
Data can be shared in consultation with the principal investigator.
Time Frame: Data can be shared after the research is published in consultation with the principal investigator.
Access Criteria: Data can be shared after the research is published in consultation with the principal investigator.